CLINICAL TRIAL: NCT04036708
Title: Caregiver Early Child Development Training for Preventing Konzo From Toxic Cassava in the Democratic Republic of Congo (DRC)
Brief Title: Caregiver Training to Prevent Konzo Disease in Children in Democratic Republic of Congo (DRC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: Institut National de Recherche Biomédicale. Kinshasa, République Démocratique du Congo (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Michael J. Boivin, Professor and Director, Psychiatry Department Research Program, Michigan State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2272; R21HD098588 (NIH)
Record Dates: First submitted 2019-07-23; First posted 2019-07-30 (Actual); Results first posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-03

CONDITIONS: Malnutrition; Manihot Species Poisoning
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MISC and WTM (Experimental): Wetting method (WTM)+ Mediational Intervention for Sensitizing Caregivers (MISC) bi-weekly for 12 months.
  Interventions: Behavioral: Wetting method (WTM); Behavioral: Mediational Intervention for Sensitizing Caregivers (MISC)
- WTM only (Active Comparator): WTM trainings only (recommended standard of care) bi-weekly for 12 months.
  Interventions: Behavioral: Wetting method (WTM)

INTERVENTIONS:
Behavioral: Wetting method (WTM) — The wetting method is an evidence-based, simple process to remove cyanogens from cassava flour. It involves teaching women to add water to cassava flour and allow it to stand for 2 h in the sun or 5 h in the shade for the hydrogen cyanide gas to escape. Colorfully illustrated and durable laminated posters depicting the WTM were distributed to participating households. Women received this training bi-weekly for 12 months.
Behavioral: Mediational Intervention for Sensitizing Caregivers (MISC) — The study team used MISC to train DRC mothers in practical day-to-day activities with their children to enhance 5 key mediational processes: 1) focusing (getting the child's attention and engaging directing them to learning experiences); 2) exciting (communicating excitement, appreciation, and affection with the learning experience); 3) expanding (making the child aware of how the learning experience transcends the present situation and can include past and future issues beyond the immediate need of the moment); 4) encouraging (emotional support to foster the child's sense of security and competence); and 5) regulating (helping to direct the child's behavior in constructive ways with a goal towards self-regulation).
  Arms: MISC and WTM

SUMMARY:
The proposed research adapted the caregiver training and child neurodevelopmental assessment capacity that the PI previously built in Uganda beginning in 2008, to a community-based intervention model for the prevention of konzo in the Democratic Republic of Congo.

DETAILED DESCRIPTION:
Early childhood (1 through 4 yrs) is a period of dramatic developmental change that can be seriously compromised by exposure to toxic cyanogenic cassava (konzo disease), with potentially great impact throughout central and western sub-Sahara Africa in regions dependent on this food staple. In the face of ongoing economic instability and nutritional, medical and educational deprivation affecting konzo at-risk communities in the Democratic Republic of Congo, no programs exist for sustaining a favorable developmental milieu for these children. By establishing the viability of caregiver training interventions to enhance functionality among caregivers and improve caregiving quality while preventing konzo, this research l can benefit tens of millions of children at-risk neurodevelopmentally; not only from poorly processed cyanogenic cassava, but also from a myriad of other non-infectious and infectious diseases.

ELIGIBILITY:
Inclusion Criteria:

* Mother with at least one child aged between 1 and 4 years
* Mother is the primary caregiver of child
* Mother is 18 years of age or older

Exclusion Criteria:

* History of brain injury (infectious, traumatic, birth) in child
* Konzo disease in any family member of household
* Epilepsy in child
* Any neurodisability in child
* Caregiver is unable to participate in the year-long training

Ages: 1 Year to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 238 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Boivin, PhD, Principal Investigator — Professor
Locations (1):
- Institute National of Research National (INRB), Kinshasa, Democratic Republic of the Congo

IPD SHARING:
Plan to Share IPD: No
The study coordinator assigns a unique identification number to each research subject at entry into the study. The first page of the risk-factor questionnaire, which contains identifying information, names and addresses, is removed after data entry and stored at the field office in a locked file dedicated to this research study. The data files will include only study numbers, which are linked through a security system to a named file maintained for the purpose of informing individuals of information pertinent to their health. The name file is only accessible to the PI Professor Michael Boivin.

REFERENCES:
- [Background] Tshala-Katumbay D, Mumba N, Okitundu L, Kazadi K, Banea M, Tylleskar T, Boivin M, Muyembe-Tamfum JJ. Cassava food toxins, konzo disease, and neurodegeneration in sub-Sahara Africans. Neurology. 2013 Mar 5;80(10):949-51. doi: 10.1212/WNL.0b013e3182840b81. PMID 23460617
- [Background] Boivin MJ, Okitundu D, Makila-Mabe B, Sombo MT, Mumba D, Sikorskii A, Mayambu B, Tshala-Katumbay D. Cognitive and motor performance in Congolese children with konzo during 4 years of follow-up: a longitudinal analysis. Lancet Glob Health. 2017 Sep;5(9):e936-e947. doi: 10.1016/S2214-109X(17)30267-X. PMID 28807191
- [Background] Boivin MJ, Okitundu D, Makila-Mabe Bumoko G, Sombo MT, Mumba D, Tylleskar T, Page CF, Tamfum Muyembe JJ, Tshala-Katumbay D. Neuropsychological effects of konzo: a neuromotor disease associated with poorly processed cassava. Pediatrics. 2013 Apr;131(4):e1231-9. doi: 10.1542/peds.2012-3011. Epub 2013 Mar 25. PMID 23530166
- [Background] Kashala-Abotnes E, Sombo MT, Okitundu DL, Kunyu M, Bumoko Makila-Mabe G, Tylleskar T, Sikorskii A, Banea JP, Mumba Ngoyi D, Tshala-Katumbay D, Boivin MJ. Dietary cyanogen exposure and early child neurodevelopment: An observational study from the Democratic Republic of Congo. PLoS One. 2018 Apr 17;13(4):e0193261. doi: 10.1371/journal.pone.0193261. eCollection 2018. PMID 29664942

RESULTS

PARTICIPANT FLOW:
Groups:
- MISC and WTM, Children; MISC and WTM, Caregivers: Wetting method (WTM)+ Mediational Intervention for Sensitizing Caregivers (MISC) bi-weekly for 12 months.
  Wetting method (WTM): The wetting method is an evidence-based, simple process to remove cyanogens from cassava flour. It involves teaching women to add water to cassava flour and allow it to stand for 2 h in the sun or 5 h in the shade for the hydrogen cyanide gas to escape. Colorfully illustrated and durable laminated posters depicting the WTM will be distributed to participating households. Women will receive this training bi-weekly for 12 months
  Mediational Intervention for Sensitizing Caregivers (MISC): The study team will use MISC to train DRC mothers in practical day-to-day activities with their children to enhance 5 key mediational processes: 1) focusing (getting the child's attention and engaging directing them to learning experiences); 2) exciting (communicating excitement, appreciation, and affection with the learning experience); 3) expanding (making the child aware of how the learning experience transcends the present situation and can include past and future issues beyond the immediate need of the moment); 4) encouraging (emotional support to foster the child's sense of security and competence); and 5) regulating (helping to direct the child's behavior in constructive ways with a goal towards self-regulation).
- WTM Only, Children; WTM Only, Caregivers: WTM trainings only (recommended standard of care) bi-weekly for 12 months.
  Wetting method (WTM): The wetting method is an evidence-based, simple process to remove cyanogens from cassava flour. It involves teaching women to add water to cassava flour and allow it to stand for 2 h in the sun or 5 h in the shade for the hydrogen cyanide gas to escape. Colorfully illustrated and durable laminated posters depicting the WTM will be distributed to participating households. Women will receive this training bi-weekly for 12 months
Period: Overall Study
Arm/Group | MISC and WTM, Children | WTM Only, Children | MISC and WTM, Caregivers | WTM Only, Caregivers
Started | 79 | 40 | 79 | 40
Completed | 65 | 36 | 65 | 36
Not Completed | 14 | 4 | 14 | 4
Not completed — Lost to Follow-up | 14 | 4 | 14 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MISC and WTM, Children | WTM Only, Children | MISC and WTM, Caregivers | WTM Only, Caregivers | Total
Number analyzed (Participants) | 79 | 40 | 79 | 40 | 238
Age, Continuous [Mean (Standard Deviation); unit: years] | 2.38 (0.68) | 2.34 (0.74) | 28.46 (8.37) | 27.98 (9.05) | 15.44 (4.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 23 | 79 | 40 | 189
  Male | 32 | 17 | 0 | 0 | 49
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 79 | 40 | 79 | 40 | 238
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Child Mullen Scales Learning Composite [Mean (Standard Deviation); unit: t-score] — The Mullen Scales of Early Learning (MSEL) assesses child developmental domains: visual reception, gross motor skills, fine motor skills, receptive language, and expressive language. A composite t-score derived from standardized t-scores of the four domains (excluding gross motor) provides a measure of g, the general measure of fluid intelligence thought to underlie general cognitive ability. The composite t-score ranges from 40 to 130. The t-scores have mean 100 and standard deviation 10 in the Western population. Higher scores reflect better outcome. Population: This measure is applicable to children only. Data were not collected from caregivers.
  t-score
    number analyzed (Participants) | 79 | 40 | 0 | 0 | 119
    (all) | 73.13 (12.09) | 74.41 (11.13) |  |  | 73.56 (11.74)
HOME score quality caregiving [Mean (Standard Deviation); unit: score on a scale] — Home Observation for the Measurement of the Environment (HOME) composite measure designed to assess the quality and quantity of stimulation that the child is exposed to in their home environment. The Infant/Toddler version includes 45 items answered on the scale from 0=none to 3=good. A total HOME score was generated by summing item responses. Potential range is 0 to 135. Higher HOME scores indicate higher quality of home environment. Population: This measure is applicable to children only. Data were not collected from caregivers.
  score on a scale
    number analyzed (Participants) | 79 | 40 | 0 | 0 | 119
    (all) | 64.88 (18.01) | 69.30 (14.59) |  |  | 66.36 (16.99)
Child Length for age z-score [Mean (Standard Deviation); unit: Z-score] — Length for age z-score was determined using the World Health Organization (WHO) algorithm using child's length, sex, and age at the time of measurement. The world population mean is 0 with standard deviation 1. Z-scores of -2 or below are often used to indicate stunting. Population: This measure is applicable to children only. Data were not collected from caregivers.
  Z-score
    number analyzed (Participants) | 79 | 40 | 0 | 0 | 119
    (all) | -1.44 (1.53) | -1.79 (1.34) |  |  | -1.56 (1.47)
Child weight-for-age z-score [Mean (Standard Deviation); unit: Z-score] — Weight for age z-score was determined using the World Health Organization (WHO) algorithm using child's length, sex, and age at the time of measurement. The world population mean is 0 with standard deviation 1. Population: This measure is applicable to children only. Data were not collected from caregivers.
  Z-score
    number analyzed (Participants) | 79 | 40 | 0 | 0 | 119
    (all) | -0.80 (1.14) | -1.23 (1.21) |  |  | -0.95 (1.17)
Bradbury Cyanide level cassava flour [Mean (Standard Deviation); unit: parts per million] — A sample of household cassava flour was collected and sent to the laboratory. Cyanide content was measured in parts per million (ppm). The WHO safe limit is 10 ppm. The range in this study was 0-200 ppm. Greater value reflects worse outcome.
  This is a household-level measure; household includes child and caregiver.
  parts per million | 28.89 (33.10) | 22.03 (24.39) | 28.89 (33.10) | 22.03 (24.39) | 26.87 (27.23)
Child urine thiocyanate [Mean (Standard Deviation); unit: Micromol per Liter] — Technicians collected samples of urine on the same day as child assessments, so that they are contiguous with level of cyanide exposure from current poorly processed cassava. Urine thiocyanite levels in urine were measured in micromol per liter. The range was 0-1032, higher scores reflect worse outcome. Population: This measure is applicable to children only. Data were not collected from caregivers.
  Micromol per Liter
    number analyzed (Participants) | 79 | 40 | 0 | 0 | 119
    (all) | 179.37 (207.35) | 227.57 (193.85) |  |  | 208.45 (202.33)
Caregiver anxiety [Mean (Standard Deviation); unit: score on a scale] — The modified Hopkins Symptom Checklist was used to assess caregiver anxiety. The instrument included 9 yes/no items, and the item responses were summed into the total score. The potential range was 0-9 with higher score indicating worse anxiety. Population: This measure is applicable to caregivers only. Data were not collected from children.
  score on a scale
    number analyzed (Participants) | 0 | 0 | 79 | 40 | 119
    (all) |  |  | 3.29 (2.96) | 3.35 (2.76) | 3.31 (2.88)
Caregiver depression [Mean (Standard Deviation); unit: score on a scale] — The modified Hopkins Symptom Checklist was used to assess caregiver depressive symptoms. The instrument included 9 yes/no items, and the item responses were summed into the total score. The potential range was 0-9 with higher score indicating worse depressive symptoms. Population: This measure is applicable to caregivers only. Data were not collected from children.
  score on a scale
    number analyzed (Participants) | 0 | 0 | 79 | 40 | 119
    (all) |  |  | 3.01 (2.37) | 2.38 (2.54) | 2.80 (2.86)

OUTCOME MEASURES:

1. Primary Outcome: Mullen Scales of Early Learning (MSEL) Composite Score
Description: The Mullen Scales of Early Learning (MSEL) assesses child developmental domains: visual reception, gross motor skills, fine motor skills, receptive language, and expressive language. A composite t-score derived from standardized t-scores of the four domains (excluding gross motor) provides a measure of g, the general measure of fluid intelligence thought to underlie general cognitive ability. The composite t-score ranges from 40 to 130. The t-scores have mean 100 and standard deviation 15 in the Western population. Higher scores reflect better outcome. Measure is applicable to children only, not collected from caregivers
Time Frame: Month 6, month 12
Population: Children
Measure: Least Squares Mean (Standard Error); unit: t-score
Arm/Group | MISC and WTM, Children | WTM Only, Children
Number analyzed (Participants) | 79 | 40
t-score
  Month 6 | 73.63 (1.33) | 74.33 (1.90)
  Month 12 | 77.04 (1.48) | 76.75 (1.93)
Statistical Analysis 1: Comparison: MISC and WTM, Children vs WTM Only, Children; The null hypothesis was that the means of two groups were equal. The alternative hypothesis was that the means of two groups were not equal. Planned sample size of total 100 analyzed was determined by feasibility considerations for this exploratory developmental R21 study. With planned n=66 in MISC+WTM arm and n=34 in WTM only arm, the unadjusted effect size of 0.60 was detectable as statistically significant with power of 0.80 and 0.05 level of significance in two-tailed tests; Test type: Superiority — The key parameter was the coefficient for the trial arm difference at month 6 in linear mixed effects model; p = .77, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. The a priori threshold for statistical significance was .05; Baseline value of the outcome, household material possessions, and the HOME score were adjusted for in the model; Mean Difference (Final Values) = 0.69, 95% CI 2-sided [-3.93 to 5.32], Standard Error of Mean 2.33 — WTM only minus MISC and WTM
Statistical Analysis 2: Comparison: MISC and WTM, Children vs WTM Only, Children; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — The key parameter was the coefficient for the trial arm difference at month 12 in linear mixed effects model; p = .90, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. The a priori threshold for statistical significance was .05; Baseline value of the outcome, household material possessions, and the HOME score were adjusted for in the model; Mean Difference (Final Values) = -0.30, 95% CI 2-sided [-5.14 to 4.54], Standard Error of Mean 2.44 — WTM only minus MISC and WTM

2. Primary Outcome: Child Urine Thiocyanite Level
Description: Technicians collected samples of urine on the same day as child assessments, so that they are contiguous with level of cyanide exposure from current poorly processed cassava. Urine thiocyanite levels in urine were measured in micromol per liter. The range was 0-1032, higher scores reflect worse outcome. Data collected from children only, not collected from caregivers.
Time Frame: Month 6, month 12
Population: Children
Measure: Least Squares Mean (Standard Error); unit: Micromol per Liter
Arm/Group | MISC and WTM, Children | WTM Only, Children
Number analyzed (Participants) | 79 | 40
Micromol per Liter
  Month 6 | 74.98 (13.94) | 139.00 (20.17)
  Month 12 | 146.45 (14.36) | 108.91 (20.18)
Statistical Analysis 1: Comparison: MISC and WTM, Children vs WTM Only, Children; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — The key parameter was the coefficient for the trial arm difference at month 6 in linear mixed effects model; p = .01, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. The a priori threshold for statistical significance was .05; Baseline value of the outcome, household material possessions, the HOME score, child's age and sex were adjusted for in the model; Mean Difference (Final Values) = 64.03, 95% CI 2-sided [15.26 to 112.8], Standard Error of Mean 24.55 — WTM only minus MISC and WTM
Statistical Analysis 2: Comparison: MISC and WTM, Children vs WTM Only, Children; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — The key parameter was the coefficient for the trial arm difference at month 12 in linear mixed effects model; p = .13, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. The a priori threshold for statistical significance was .05; Baseline value of the outcome, household material possessions, the HOME score, and child's age and sex were adjusted for in the model; Mean Difference (Final Values) = -37.53, 95% CI 2-sided [-86.92 to 11.85], Standard Error of Mean 24.86 — WTM only minus MISC and WTM

3. Secondary Outcome: Home Observation for the Measurement of the Environment (HOME) Score
Description: Home Observation for the Measurement of the Environment (HOME) composite measure designed to assess the quality and quantity of stimulation that the child is exposed to in their home environment. The Infant/Toddler version includes 45 items answered on the scale from 0=none to 3=good. A total HOME score was generated by summing item responses. Potential range is 0 to 135. Higher HOME scores indicate higher quality of home environment. Measure applies to children only.
Time Frame: Month 6, month 12
Population: Children
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | MISC and WTM, Children | WTM Only, Children
Number analyzed (Participants) | 79 | 40
score on a scale
  Month 6 | 69.37 (1.70) | 67.61 (2.42)
  Month 12 | 71.49 (1.84) | 68.07 (2.42)
Statistical Analysis 1: Comparison: MISC and WTM, Children vs WTM Only, Children; The null hypothesis was that the means of two groups were equal. Sample size was determined by considerations for the primary outcomes; Test type: Superiority — The key parameter was the coefficient for the trial arm difference at month 6 in linear mixed effects model; p = .55, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. The a priori threshold for statistical significance was .05; Baseline value of the outcome and household material possessions were adjusted for in the model; Mean Difference (Final Values) = -1.76, 95% CI 2-sided [-7.65 to 4.13], Standard Error of Mean 2.97 — WTM only minus MISC and WTM
Statistical Analysis 2: Comparison: MISC and WTM, Children vs WTM Only, Children; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — The key parameter was the coefficient for the trial arm difference at month 12 in linear mixed effects model; p = .26, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. The a priori threshold for statistical significance was .05; Baseline value of the outcome and household material possessions were adjusted for in the model; Mean Difference (Final Values) = -3.42, 95% CI 2-sided [-9.48 to 2.63], Standard Error of Mean 3.05 — WTM only minus MISC and WTM

4. Secondary Outcome: Child Physical Growth: Length for Age Z-score
Description: Length for age z-score was determined using the World Health Organization algorithm using child's length, sex, and age at the time of measurement. The world population mean is 0 with standard deviation 1. Z-scores of -2 or below are often used to indicate stunting.
Time Frame: Month 6, month 12
Population: Children
Measure: Least Squares Mean (Standard Error); unit: z-score
Arm/Group | MISC and WTM, Children | WTM Only, Children
Number analyzed (Participants) | 79 | 40
z-score
  Month 6 | -1.72 (0.09) | -1.88 (0.13)
  Month 12 | -1.57 (0.10) | -1.96 (0.13)
Statistical Analysis 1: Comparison: MISC and WTM, Children vs WTM Only, Children; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — The key parameter was the coefficient for the trial arm difference at month 6 in linear mixed effects model; p = .32, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. The a priori threshold for statistical significance was .05; Baseline value of the outcome, household material possessions, and the HOME score were adjusted for in the model; Mean Difference (Final Values) = -0.16, 95% CI 2-sided [-0.48 to 0.16], Standard Error of Mean 0.16 — WTM only minus MISC and WTM
Statistical Analysis 2: Comparison: MISC and WTM, Children vs WTM Only, Children; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — The key parameter was the coefficient for the trial arm difference at month 12 in linear mixed effects model; p = .02, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. The a priori threshold for statistical significance was .05; Baseline value of the outcome, household material possessions, and the HOME score were adjusted for in the model; Mean Difference (Final Values) = -0.39, 95% CI 2-sided [-0.72 to -0.06], Standard Error of Mean 0.16 — WTM only minus MISC and WTM

5. Secondary Outcome: Child Physical Growth: Weight for Age Z-score
Description: Weight for age z-score was determined using the World Health Organization algorithm using child's length, sex, and age at the time of measurement. The world population mean is 0 with standard deviation 1.
Time Frame: Month 6, month 12
Population: Children
Measure: Least Squares Mean (Standard Error); unit: z-score
Arm/Group | MISC and WTM, Children | WTM Only, Children
Number analyzed (Participants) | 79 | 40
z-score
  Month 6 | -1.54 (0.12) | -1.92 (0.16)
  Month 12 | -1.40 (0.13) | -2.10 (0.16)
Statistical Analysis 1: Comparison: MISC and WTM, Children vs WTM Only, Children; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — The key parameter was the coefficient for the trial arm difference at month 6 in linear mixed effects model; p = .06, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. The a priori threshold for statistical significance was .05; Baseline value of the outcome, household material possessions, and the HOME score were adjusted for in the model; Mean Difference (Final Values) = -0.38, 95% CI 2-sided [-0.78 to 0.01], Standard Error of Mean 0.20 — WTM only minus MISC and WTM
Statistical Analysis 2: Comparison: MISC and WTM, Children vs WTM Only, Children; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — The key parameter was the coefficient for the trial arm difference at month 12 in linear mixed effects model; p = .001, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. The a priori threshold for statistical significance was .05; Baseline value of the outcome, household material possessions, and the HOME score were adjusted for in the model; Mean Difference (Final Values) = -0.70, 95% CI 2-sided [-1.11 to -0.28], Standard Error of Mean 0.21 — WTM only minus MISC and WTM

6. Secondary Outcome: Caregiver Anxiety Symptoms
Description: The modified Hopkins Symptom Checklist was used to assess caregiver anxiety. The instrument included 9 yes/no items, and the item responses were summed into the total score. The potential range was 0-9 with higher score indicating worse anxiety. Measure applicable to caregiver only. Data were not collected from children.
Time Frame: Month 6, month 12
Population: Caregivers of children
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | MISC and WTM, Caregivers | WTM Only, Caregivers
Number analyzed (Participants) | 79 | 40
score on a scale
  Month 6 | 2.86 (0.28) | 3.91 (0.40)
  Month 12 | 2.80 (0.30) | 3.74 (0.41)
Statistical Analysis 1: Comparison: MISC and WTM, Caregivers vs WTM Only, Caregivers; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — The key parameter was the coefficient for the trial arm difference at month 6 in linear mixed effects model; p = .04, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. The a priori threshold for statistical significance was .05; Baseline value of the outcome, household material possessions, and the HOME score were adjusted for in the model; Mean Difference (Final Values) = 1.05, 95% CI 2-sided [0.07 to 2.03], Standard Error of Mean 0.49 — WTM only minus MISC and WTM
Statistical Analysis 2: Comparison: MISC and WTM, Caregivers vs WTM Only, Caregivers; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — The key parameter was the coefficient for the trial arm difference at month 12 in linear mixed effects model; p = .07, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. The a priori threshold for statistical significance was .05; Baseline value of the outcome, household material possessions, and the HOME score were adjusted for in the model; Mean Difference (Final Values) = 0.94, 95% CI 2-sided [-0.08 to 1.96], Standard Error of Mean 0.51 — WTM only minus MISC and WTM

7. Secondary Outcome: Caregiver Depressive Symptoms
Description: The modified Hopkins Symptom Checklist was used to assess caregiver depressive symptoms. The instrument included 9 yes/no items, and the item responses were summed into the total score. The potential range was 0-9 with higher score indicating worse depressive symptoms. Measure applies to caregivers only, data were not collected from children.
Time Frame: Month 6, month 12
Population: Caregivers of children
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | MISC and WTM, Caregivers | WTM Only, Caregivers
Number analyzed (Participants) | 79 | 40
score on a scale
  Month 6 | 2.21 (0.29) | 4.25 (0.42)
  Month 12 | 2.45 (0.32) | 4.18 (0.42)
Statistical Analysis 1: Comparison: MISC and WTM, Caregivers vs WTM Only, Caregivers; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — The key parameter was the coefficient for the trial arm difference at month 6 in linear mixed effects model; p < .01, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. The a priori threshold for statistical significance was .05; Baseline value of the outcome, household material possessions, and the HOME score were adjusted for in the model; Mean Difference (Final Values) = 2.04, 95% CI 2-sided [1.02 to 3.06], Standard Error of Mean 0.51 — WTM only minus MISC and WTM
Statistical Analysis 2: Comparison: MISC and WTM, Caregivers vs WTM Only, Caregivers; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — The key parameter was the coefficient for the trial arm difference at month 12 in linear mixed effects model; p < .01, Mixed Models Analysis — P-value was not adjusted for multiple comparisons. The a priori threshold for statistical significance was .05; Baseline value of the outcome, household material possessions, and the HOME score were adjusted for in the model; Mean Difference (Final Values) = 1.73, 95% CI 2-sided [0.67 to 2.79], Standard Error of Mean 0.53 — WTM only minus MISC and WTM

ADVERSE EVENTS:
Time Frame: 12 months after enrollment into the study
Description: Adverse events were determined as part of study assessments at months 6 and 12.
Groups:
- MISC and WTM, Children; MISC and WTM, Caregivers: Wetting method (WTM)+ Mediational Intervention for Sensitizing Caregivers (MISC) bi-weekly for 12 months.
  Wetting method (WTM): The wetting method is an evidence-based, simple process to remove cyanogens from cassava flour. It involves teaching women to add water to cassava flour and allow it to stand for 2 h in the sun or 5 h in the shade for the hydrogen cyanide gas to escape. Colorfully illustrated and durable laminated posters depicting the WTM were distributed to participating households. Women received this training bi-weekly for 12 months.
  Mediational Intervention for Sensitizing Caregivers (MISC): The study team used MISC to train DRC mothers in practical day-to-day activities with their children to enhance 5 key mediational processes: 1) focusing (getting the child's attention and engaging directing them to learning experiences); 2) exciting (communicating excitement, appreciation, and affection with the learning experience); 3) expanding (making the child aware of how the learning experience transcends the present situation and can include past and future issues beyond the immediate need of the moment); 4) encouraging (emotional support to foster the child's sense of security and competence); and 5) regulating (helping to direct the child's behavior in constructive ways with a goal towards self-regulation).
- WTM Only, Children; WTM Only, Caregivers: WTM trainings only (recommended standard of care) bi-weekly for 12 months.
  Wetting method (WTM): The wetting method is an evidence-based, simple process to remove cyanogens from cassava flour. It involves teaching women to add water to cassava flour and allow it to stand for 2 h in the sun or 5 h in the shade for the hydrogen cyanide gas to escape. Colorfully illustrated and durable laminated posters depicting the WTM were distributed to participating households. Women received this training bi-weekly for 12 months.
Arm/Group | MISC and WTM, Children | WTM Only, Children | MISC and WTM, Caregivers | WTM Only, Caregivers
All-Cause Mortality (participants affected / at risk) | 0/79 | 0/40 | 0/79 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/79 | 0/40 | 0/79 | 0/40
Other Adverse Events (participants affected / at risk) | 0/79 | 0/40 | 0/79 | 0/40

LIMITATIONS AND CAVEATS:
The study was exploratory and developmental in nature. Where statistical significance was not reached, estimates of the means and standard deviations will be used to formally power future trials of MISC and WTM interventions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-14): https://cdn.clinicaltrials.gov/large-docs/08/NCT04036708/Prot_SAP_000.pdf